CLINICAL TRIAL: NCT04384939
Title: Feasibility, Safety and Medico-economic Study of Magnetic-end Double-J Ureteral Stent Use in Children
Brief Title: Feasibility of Magnetic-end Double-J Ureteral Stent Use in Children
Acronym: EFUJA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP180426; 2018-A0295550 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-02-20; First posted 2020-05-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Uropathy; Kidney Transplantation
Keywords: Double-J ureteral stent (DJUS); magnetic-end; Pediatric urology; Uropathy; Kidney graft
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Double-J ureteral stent (Experimental): Pediatric patient with an uropathy or kidney graft need the insertion of Double-J ureteral stent in a routine care
  Interventions: Device: magnetic-end Double-J ureteral stent

INTERVENTIONS:
Device: magnetic-end Double-J ureteral stent — * Inserting the ureteral stent with magnet (same process as classic ureteral stent)
  * Removing the ureteral stent with magnet without general anaesthesia. Usually, the classic ureteral stent removed during a general anaesthesia.
  Other Names: No applied

SUMMARY:
Double-J ureteral stent (DJUS) is one of the most common devices used in urology. Ureteral stenting has a wide spectrum of indications that can be summarized in two words: obstruction and leakage. Common indications in pediatric urology are pyeloplasty, ureteral reimplantation, kidney transplantation and stone disease.

Classically, DJUS are introduced and removed in the operation room, under general anesthesia, using a cystoscope.

The magnetic-end Double-J ureteral stent is a 4.8 French DJUS with a small magnet fixed with a string at the distal loop.

To remove the magnetic stent, a 9 French customized catheter-like retrieval device with a magnetic Tiemann tip is inserted into the urethra in the outpatient clinic.

The purpose of this study is to demonstrate the feasibility and safety of magnetic-end Double-J ureteral stent use in children and to perform a medico-economic study.

DETAILED DESCRIPTION:
First reported in 1967, ureteral stenting evolved fast until the introduction of the double-J ureteral stent (DJUS) in 1978. It has since become one of the most common devices used in urology. Ureteral stenting has a wide spectrum of indications that can be summarized in two words: obstruction and leakage. Common indications in pediatric urology are pyeloplasty, ureteral reimplantation, kidney transplantation and stone disease.

Many modifications have been introduced to Finney's double-J to reduce stent-related complications and disadvantages, one of which is its removal technique. Classically, DJUS are introduced and removed in the operation room (OR), under general anesthesia (GA), using a cystoscope. Efforts have been made to avoid the second procedure under GA. Preventing the patient from undergoing a second OR experience is not the only issue. For institutions, DJUS removal is time consuming and costly in terms of resources, OR occupancy, and staff. In children, the potential neurotoxicity of repeated exposures to GA, is also a major concern.

Alternatives to surgical removal of DJUS vary from basic solutions such as transurethral string, hook, or other tools, to more complex innovations such as the single use flexible cystoscope, and biodegradable stents. Moreover, some pediatric teams used the externalized pyeloureteral stent as an alternative to DJUS. Using magnet for ureteral stent retrieval was introduced in the early 80s. Difficulties related to its insertion, as well as its low retrieval success rate, minimized its acceptance. It wasn't until 2002 when Taylor and McDougall revisited the concept of magnetic retrieval of the ureteral stent. Since then, few teams have published their experience with magnetic-end DJUS.

The magnetic-end Double-J ureteral stent is a 4.8 French DJUS with a small magnet fixed with a string at the distal loop. Explanation of the retrieval method and its potential complications are given to the parents, and informed consent obtained prior to surgery. All of the stents are inserted under GA in the exact same manner as regular DJUS: antegrade, retrograde (cystoscopy insertion) or open surgery. The stent's length varies between 12 and 24 cm depending on the age and weight of the child. An abdominal plain X-Ray is routinely done after pyeloplasty to check the position of the DJUS distal loop (MEDJUS or not) in the bladder before waking up the child. A successful stent insertion is defined as having a good position of the distal end and its magnet in the bladder

To remove the magnetic-end Double-J ureteral stent, a 9 French customized catheter-like retrieval device with a magnetic Tiemann tip, lubricated with 2% lidocaine jelly, is inserted into the urethra by the surgeon with the patient breathing inhaled premixed nitrous oxide and oxygen for procedural sedation in the outpatient clinic. Both indwelling magnets connect and the catheter can be removed together with the MEDJUS. Success of magnetic retrieval are regarded as MEDJUS retrieval in outpatient clinic with no need of general anesthesia.

The aim is to demonstrate the feasibility and safety of the magnetic-end DJUS in children and perform a medico-economic study / cost-effectiveness study to evaluate the impact of the use of MEDJUS in children in terms of retrieval time and cost, as well as OR and staff occupancy.

ELIGIBILITY:
Inclusion Criteria:

* Child aged between 0 and 17 years and 10 months at the surgery
* Child operated at the Necker hospital for an uropathy or kidney graft need the insertion of JJ ureteral stent
* Parents or legal guardians signed the Informed consent form
* Social insurance affiliation

Exclusion Criteria:

* All clinical situation need an MRI
* Contraindication with the experimental medical device (severe infections, obstruction, …)

For the medico-economic study, a comparative group will be constituted with patients treated with classic ureteral stent in the Necker hospital in the previous years.

This group will be matched with age (<5 years, 5-12 years and >13years), sex and surgery indication (kidney graft or other).

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Successful removal of the Double-J ureteral stent with magnet | During the stent removal consultation, usually between 8 and 30 days after the surgery
  A successful removal is a removal of the Double-J (JJ) ureteral stent with the magnet removal system, without general anaesthesia - The measure is a binary criterion: success/ failure, evaluated by the surgeon

SECONDARY OUTCOMES:
Successful insertion of the Double-J ureteral stent with magnet | 1 day
  A successful insertion is an insertion of the JJ ureteral stent with magnet in retrograde, antegrade process or open surgery - The measure is a binary criterion: success/ failure, evaluated by the surgeon
Duration of hospitalization | At the end of the initial hospitalisation, at maximum 60 days
  Number of total days of hospitalization
Costs of hospitalization after surgery | Until the stent removal consultation, usually between 8 and 30 days after the surgery
  Costs of hospitalization after surgery
Pain score | At the end of the stent removal
  EVA or EVENDOL pain assessment on the child's age prior to, during, and subsequent to the removal
Anxiety score | At the end of the stent removal
  Anxiety assessment using the mYPAS scale (modified-Yale Preoperative Anxiety Scale) consisting of 27 items divided into 5 categories: Activity, Vocalizations, Emotional Expressivity, State of Arousal and Use of Parent.- higher score indicating higher anxiety
Satisfaction survey of parents | at the end of the stent removal and day 7 after
  A satisfaction survey that parents completed on D7 and at the end of the stent removal

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BLANC, MD, PhD, Principal Investigator — Assistance Publique -Hôpitaux de Paris (AP-HP)
Locations (1):
- Hôpital Necker, Paris, France